CLINICAL TRIAL: NCT05199493
Title: Biomarker-guided Implementation of Angiotensin-II (AT-II) to Reduce the Occurrence of Kidney Damage After Cardiac Surgery
Brief Title: Reducing Acute Kidney Injury Occurence by Administering Angiotensin II
Acronym: AIDED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universität Münster (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WWU20_0016; 2021-003088-87 (EudraCT Number); 06-AnIt-20 (Other: Dept. of Anesthesiology, Intensive Care and Pain Medicine)
Record Dates: First submitted 2021-12-02; First posted 2022-01-20 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Cardiac Surgery; Vasoplegia; Hyperreninemia
Keywords: Cardiac Surgery; Acute kidney injury; Biomarker; Angiotensin II; Renin
MeSH Terms: conditions — Vasoplegia; Acute Kidney Injury | interventions — Angiotensin II

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiotensin II (Experimental): Intravenous infusion of max. 80 ng/kg/min Angiotensin II (titrated for each individual patient by effect) over 12 h after start of infusion
  Interventions: Drug: Angiotensin II
- Control (Placebo Comparator): Intravenous infusion placebo (matched infusion volume) over 12 h after start of infusion
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Angiotensin II — Patients with Delta-renin >= 3.7 micro-unit/mL are at high risk for AKI. Patients who have a high delta-renin and a postoperative hypotension requiring vasopressors ad will be randomized. After randomization patients will receive intravenous infusion with the investigational drug.
  Arms: Angiotensin II
Drug: Control — Patients with Delta-renin >= 3.7 micro-unit/mL are at high risk for AKI. Patients who have a high delta-renin and a postoperative hypotension requiring vasopressors ad will be randomized. After randomization patients will receive intravenous infusion with placebo
  Arms: Control

SUMMARY:
The aim of this study is to evaluate whether adding angiotensin II to the standard of care is superior compared to the standard of care alone with respect to kidney damage (personalized approach) after cardiac surgery.

DETAILED DESCRIPTION:
Vasoplegic syndrome is a form of distributive shock that is characterized by low arterial pressure with reduced systemic vascular resistance and normal or elevated cardiac output that occurs in 5 to 25% of patients undergoing cardiac surgery. Patients with vasoplegic shock after cardiac surgery are at higher risk of organ failure, including acute kidney injury (AKI). Postsurgical AKI is associated with several adverse outcomes. Attempts to prevent AKI have largely been futile so far. Prior studies often started with the interventions after an AKI event, when a decline of kidney function (i.e. glomerular filtration rate) was already established. Application of norepinephrine is currently considered as the first-line therapy for vasoplegic shock, but all catecholamines have adverse effects, including myocardial ischemia and arrhythmias. In a recent observational trial, we demonstrated that there is a dysregulation in the renin-angiotensin-aldosterone system (RAAS) likely caused by a reduced angiotensin-converting enzyme (ACE) activity after cardiac surgery. Elevated renin levels identified patients at risk for AKI and were associated with cardiovascular instability and increased AKI rate after cardiac surgery. Furthermore, elevated renin levels could be used to identify high-risk patients for cardiovascular instability and AKI who would benefit from timely intervention with angiotensin II that could improve their outcomes. Therefore, the application of angiotensin II to treat a postoperative hypotension would mean a hormone substitution.Shock after cardiac surgery is associated with increased mortality. Cardiopulmonary bypass (CPB) represents a common clinical setting of sympathetic nervous system activation and cardiovascular instability. Vasoplegia is a form of distributive shock that is characterized by low arterial pressure with reduced systemic vascular resistance and normal or elevated cardiac output. It occurs in 5 to 25% of patients undergoing cardiac surgery. Patients with vasoplegia after cardiac surgery are at higher risk of organ failure, including AKI, and have an increased mortality rate and longer hospital length of stay.

Clinical trials focusing on septic patients suggest that AT-II is a potent vasopressor. However, no human data exist whether the application of AT-II in cardiac surgery patients with y hyperreninemia high-risk patients identified by renin levels (individualized approach) reduces kidney damage and improves kidney function after cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery with CPB
* Cardiac index 2.1l/min per square meter
* Written informed consent
* D-renin (difference between post- and preoperative) ≥ 3.7 micro Unit/ml 4 h after CPB
* Postoperative hypotension requiring vasopressors

Exclusion Criteria:

* Preexisting AKI (stage 1 and higher)
* Patients with cardiac assist devices
* Pregnant women, nursing women and women of childbearing potential
* Known (Glomerulo-) Nephritis, interstitial nephritis or vasculitis
* chronic kidney disease with estimated glomerular filtration rate (eGFR) < 30 ml/min
* Dialysis dependent chronic kidney disease
* Prior kidney transplant within the last to 12 months
* Emergency surgery in the context of an acute coronary syndrome
* Hypersensitivity to the active substance, or to any of the excipients of the study medication
* Bronchospasm
* Liver failure
* Mesenteric ischemia
* Participation in another intervention trial in the past 3 months
* Persons with any kind of dependency on the investigator or employed by the institution responsible or investigator
* Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-03-19 (Actual)

PRIMARY OUTCOMES:
• kidney damage after cardiac surgery identified by the difference between [TIMP-2]*[IGFBP7] levels 12h after randomization and [TIMP-2]*[IGFBP7] levels at randomization | 12 hours after start of intervention
  The presence of tissue inhibitor of metalloproteinases (TIMP-2) and insulin-like growth-factor binding protein 7 (IGFBP7) in the urine will be measured.

SECONDARY OUTCOMES:
Occurence of Acute Kidney Injury (AKI) according to the Kidney Disease: Improving Global Outcomes (KDIGO) criteria | 72 hours after cardiac surgery
Severity of Acute Kidney Injury | 72 hours after cardiac surgery
  Number of patients with KDIGO stage 1, KDIGO stage 2 or KDIGO stage 3)
Amount of volume application | 12 hours after start of intervention
Fluid status | 12 hours after start of intervention
Dose of vasopressor use during intervention | During intervention, an average of 12 hours
Creatinine clearance on day one after cardiac surgery | One day after cardiac surgery
Free-days through day 28 of vasoactive medications and mechanical ventilation | 28 days after cardiac surgery
Renal Recovery | 90 days after cardiac surgery
  Renal recovery is defined as serum creatinine levels < 0.5 mg/dL higher than baseline serum creatinine
Mortality | 30 days after cardiac surgery
Mortality | 60 days after cardiac surgery
Mortality | 90 days after cardiac surgery
Length of ICU (Intensive Care Unit) stay | up to 90 days after cardiac surgery (until discharge)
Length of hospital stay | up to 90 days after cardiac surgery (until discharge)
Use and duration of renal replacement therapy | up to 90 days after cardiac surgery
  Number of patients with renal replacement therapy
Major adverse kidney events (MAKE) | 90 days after cardiac surgery
  Major adverse kidney events consisting of mortality, dialysis dependency, persistent renal dysfunction (defined as serum creatinine ≥ 2x compared to baseline value)
Effect of Angiotensin converting enzyme inhibitor (ACEi)/angiotensin II receptor blocker (ARBs) use on the effect of angiotensin II | 12 hours after intervention
Correlation between the severity of hyperreninemia and the effect of angiotensin II | 12 hours after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zarbock, MD, Study Chair — University Hospital Muenster, Dept. of Anesthesiology, Intensive Care Medicine and Pain Therapy
Locations (1):
- University Hospital Muenster, Münster, Germany

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT05199493/Prot_000.pdf